CLINICAL TRIAL: NCT02361099
Title: Phase 3 Multicentric Randomized Study Assessing Self-reported Symptoms Transmitted Via an Internet Web-application " Sentinel " Versus Conventional Follow-up in Patients With High Risk Lung Cancer (SENTINEL)
Brief Title: SENTINEL : Impact of the Use of a Web-application for the Detection of Lung Cancer Relapse
Acronym: SENTINEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weprom (Other)
Collaborators: Sivan Innovation Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WP-2018-01; 2014-A00263-44 (Other: RCB)
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitoring by SENTINEL application (Experimental): Patients randomized to this arm will connect once a week to SENTINEL application to do a self-evaluation of several symptoms. A CT- scan will be scheduled only when there is an alert of the application.
  Interventions: Other: Monitoring by SENTINEL application
- Conventional Monitoring (No Intervention): Patients randomized to this arm will have a CT-scan every 3 months.

INTERVENTIONS:
Other: Monitoring by SENTINEL application — Patients will connect once a week to SENTINEL application to do a self-evaluation of several symptoms. A CT- scan will be scheduled only when there is an alert of the application
  Other Names: new technology
  Arms: Monitoring by SENTINEL application

SUMMARY:
This is a study that evaluates an optimization of the monitoring of patients with lung cancer in order to extend the survival of patients by improving their quality of life and decreasing anxiety generated by the achievement of balance sheets imaging. The spacing of the follow-up imaging also helps to reduce the cost of such monitoring. The main objective of this study is to evaluate the overall survival of patients.

DETAILED DESCRIPTION:
With a 5-year survival of about 15% pulmonary cancer is very poor prognosis. About 70 to 75% of cancers are diagnosed at advanced stages. Relapses are common and rarely curable. At least 75% of relapses are symptomatic and there is no standard monitoring after curative treatment or not. Currently, the most common monitoring strategy involves the completion of a clinical examination every 3 to 6 months associated with chest X-ray or CT-scan.

An intensive clinical and imaging monitoring has not yet shown any survival advantage but monitoring of symptoms appears to have a significant medical and economic advantage compared to imaging monitoring. This non-personalized approach is a source of anxiety for patients, especially with the approach of the date of the imaging assessment. In contrast, this monitoring can leave symptomatic patients with untreated relapse for several weeks because many symptomatic patients wait the date of the imaging assessment to consult.

the investigators have developed a score based on the dynamics and the association of clinical signs to alert the physician to a possible recurrence of lung cancer. The referring physician is alerted so early and convenes the patient for a checkup. One of the explanations which could demonstrate the gain in survival is the possibility offered by the application SENTINEL is to treat the relapses earlier, thus avoiding to wait a too much important deterioration of general condition between two monitoring follow-up more or less spaced.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with lung cancer (NSCLC and SCLC), histologically proven
2. Patient at high risk of relapse (TxN1, IIIA, IIIB, IV stages)
3. Age ≥ 18 ans
4. PS ≤ 2 within 15 days before enrollment
5. Patient having:

   * finished his cancer treatment in the last 3 months by:

     * Surgery or
     * Surgery then adjuvant chemotherapy or
     * Concomitant radio-chemotherapy or
     * Conventional or stereotactic radiotherapy or
     * 1st or 2nd line chemotherapy
   * treatment with TKI (tyrosine kinase inhibitor) in 1st or 2nd line or maintenance treatment with Alimta® and / or Avastin® or Gemzar® well tolerated (SENTINEL 's score with this treatment (TKI or maintenance) to its latest assessment.
6. Patient with an initial SENTINEL score ≤ 6
7. Patient with internet access and an e-mail box
8. Patient affiliated to a social security scheme
9. Patient has given its written consent before any specific procedure from protocol

Exclusion Criteria:

1. Patient whose disease has progressed at the end of the specific treatment
2. Symptomatic brain metastases
3. Persons deprived of liberty or under guardianship or curators
4. Dementia, mental alteration or psychiatric pathology that can compromise informed consent from the patient and / or adherence to the protocol and the monitoring of the trial
5. Patient who cannot submit himself to the followed of the protocol for psychological reasons, social, family or geographical
6. Pregnant or breastfeeding women
7. Patient participating in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 24 months
  Overall survival is defined as the period between the date of randomization to the date of death from any cause. We will also evaluate in this context the overall survival defined between the date of diagnosis and date of death whatever the cause in order to know more precisely the duration of the disease.

SECONDARY OUTCOMES:
Quality of Life (QOL) | 12 month
  The quality of life will be studied using the questionnaire FACT-L at baseline and follow-up visits at 3, 6 and 12 months.
Depression | 12 month
  Patient's depression will be assessed through the questionnaire HUMEUR PHQ9 at baseline and follow-ups at 3, 6 and 12 months.
Relapse detection time | 24 month
  The relapse detection time is defined as time from the date of diagnosis to the date of highlighting of the recurrence by imaging
Performance Status (PS) | 24 month
  Performance Status will be evaluated according to WHO recommendations.
Cost of monitoring | 24 month
  The cost of monitoring will be evaluated from the perspective of health insurance.
Patient compliance | 24 month
  Patient compliance to the use of SENTINEL application will be evaluated according to the number of assessments completed (usually 1 per week) compared to the theoretical maximum number filling weekly and monthly the application over time.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, MD, Principal Investigator — Centre Jean Bernard - LE MANS
Locations (9):
- France (9):
  - Centre Hospitalier Universitaire, Angers
  - Institut de Cancerologie de l'Ouest - site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Général, Chartres
  - Centre Hospitalier Départemenal, La Roche-sur-Yon
  - Centre Jean Bernard, Le Mans
  - Centre Hospitalier, Le Mans
  - Centre Catherine de Sienne, Nantes
  - Institut de Cancerologie de l'Ouest - site René Gauducheau, Saint-Herblain